CLINICAL TRIAL: NCT06200493
Title: Investigation of Maximum Strength and Acceleration Ability as a Function of Grip Position and Its Effects on Performance and Training in Wheelchair Sports
Brief Title: Effects of Maximum Strength and Acceleration Ability on Performance and Training in Wheelchair Sports
Acronym: OPM
Status: Completed | Type: Observational
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Other Study IDs: 2023-10
Record Dates: First submitted 2023-12-01; First posted 2024-01-11 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Spinal Cord Injuries; Athletes; Wheelchair
Keywords: maximal strength; sprint time; maximal acceleration
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Wheelchair Athletes: national squad athletes in either wheelchair rugby or wheelchair basketball

SUMMARY:
The goal of this observational study is to learn about the relation between grip position and maximal strength and power in wheelchair rugby and basketball athletes. The main question is to investigate the relationship between maximal isometric force, acceleration, and sprint time.

Participants will

* pull in their sport wheelchair against a force transducer
* push in their sport wheelchair from a force transducer
* accelerate as fast as possible with one push
* accelerate as fast as possible over a distance of 20m

Researchers will compare the wheelchair basketball against wheelchair rugby players to see if there is a difference in the parameters.

DETAILED DESCRIPTION:
The study duration is approximately 2 hours per participant. First, the screening will be done and the participant does a warmup (~30 min). After that, the participant gets ready for testing, which will last for approximately 90 minutes. In each test, the participants have trial rounds to familiarize with the test procedure. The testing consist of three different exercises, the isometric strength test (IsoMST), the maximum initial push propulsion (MIPP) and the sprint. In the IsoMST a pull setup which was already used in literature and a push setup which has yet to be validated will be used. For the pull setup, the chair of the athlete is fixated on the wall which results in a static situation and allows for an isometric effort. For the push setup, a bumper is installed on the wall, against which the athletes can push with their chair. Different grip position will be measured. In the MIPP test the participants are instructed to accelerate as quickly as possible from standstill with only one push on the rim. The MIPP will be executed with several different grip positions, equal to the IsoMST. For the sprint, 20m will be marked out on a playing court. The athletes are instructed to complete the distance as quickly as possible. Several split times as well as the total time will be measured.

ELIGIBILITY:
Inclusion Criteria:

* squad members or doing more than 3h per week wheelchair basket/rugby training
* adequately informed and consent confirmed per signature

Exclusion Criteria:

* Pregnancy based on anamnesis
* acute illness, injury, infection, etc., which would impact the measurements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: wheelchair athletes that are squad members in either wheelchair rugby or wheelchair basketball or doing more than 3h wheelchair basket/rugby training per week
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
maximal pull force | during 1 second of maximal pulling
  The maximal isometric force produced during pulling in the sport wheelchair

SECONDARY OUTCOMES:
maximal push force | during the first second of maximal pushing
  The maximal isometric force produced during pushing in the sport wheelchair
maximal acceleration | during the first second of acceleration
  The maximal acceleration reached with one push in the sport wheelchair
sprint time | during the last second of the 20 metre sprint
  The time for the linear sprint over 20m in the sport wheelchair

OTHER OUTCOMES:
rate of force development | during the first second of maximal push
  The rate of force development (RFD) in the isometric push and pull test
sprint distance time | during 5 seconds of the linear sprint
  The time for the linear sprint over sub distance in the sport wheelchair
one push maximal speed | during the last second of acceleration
  The maximal speed reached with one push in the sport wheelchair

CONTACTS AND LOCATIONS:
Locations (1):
- Swiss Paraplegic Centre, Nottwil, Canton of Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No